CLINICAL TRIAL: NCT04153669
Title: Effects of Exercise With or Without Electrical Stimulation in Physical Fitness in Cystic Fibrosis: an Integrated Vision (ECOMIRIN Study)
Brief Title: Exercise With or Without Electrical Stimulation in Cystic Fibrosis (Part I): Effects on Physical Fitness
Acronym: ECOMIRIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Margarita Perez, Full Professor in Exercise Physiology, MD, PhD, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-0019/18
Record Dates: First submitted 2019-10-30; First posted 2019-11-06 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis in Children
Keywords: Cystic Fibrosis; Electrostimulation; Combined Training; Physical Fitness
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): This group will continue with regular visits to the specialist. This visits include recommendations to improve lifestyle.
- Exercise-No NMES (Experimental): This group will continue with regular visits to the specialist. This visits include recommendations to improve lifestyle.
  The exercise protocol includes a concurrent exercise intervention (strength training and aerobic training), 3 days a week, 60 minutes sessions.
  Interventions: Behavioral: Exercise-No NMES
- Exercise-NMES (Experimental): This group will continue with regular visits to the specialist. This visits include recommendations to improve lifestyle.
  The exercise protocol includes a concurrent exercise intervention (strength training and aerobic training), 3 days a week, 60 minutes sessions. Additionally, this group will receive neuromuscular electrical stimulation (NMES) concomitant to the strength training.
  Interventions: Behavioral: Exercise-NMES

INTERVENTIONS:
Behavioral: Exercise-NMES — Exercise-NMES
  Arms: Exercise-NMES
Behavioral: Exercise-No NMES — Exercise-No NMES
  Arms: Exercise-No NMES

SUMMARY:
This study aims to assess the effects of programmed exercise with or without electrical stimulation in the cardiorespiratory fitness, strength, functional capacity and agility in a group of young patients with Cystic Fibrosis: A randomized controlled trial comparing two interventions with a control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF
* Age: 6-18 years old
* Signature of informed consent of legal guardian and patient.

Exclusion Criteria:

* Being a smoker
* Having had an exacerbation in the last 3 months
* Having undergone gastric surgery
* Having enteral nutrition at present
* The patients will come from the HIUNJ of Madrid.
* Currently taking CFTR modulators

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Change in Strength | Two assessment points throughout the study: baseline and 8 weeks after the intervention
  Changes in strength will be measured using a five repetition maximum test (5RM)

SECONDARY OUTCOMES:
Change in Cardiorespiratory Fitness | Two assessment points throughout the study:baseline and 8 weeks after the intervention
  Changes in cardiorespiratory fitness will be measured using a cardiopulmonary exercise test (CPET)
Changes in Pulmonary Function | Two assessment points throughout the study:baseline and 8 weeks after the intervention
  Changes in pulmonary function will be measured using Spirometry
Changes in physical activity levels | Two assessment points throughout the study:baseline and 8 weeks after the intervention
  Changes in physical activity levels will be measured using Physical Activity Questionnaire for Children and Adolescents (PAC-C or PAC-A)
Change in quality of life | Two assessment points throughout the study:baseline and 8 weeks after the intervention
  Changes in quality of life will be measures with the Cystic Fibrosis-Questionnaire-Revised (CFQ-R)
Food consumption frequency | One assessment point at baseline:baseline and 8 weeks after the intervention
  The food consumption frequency will be measured using food frequency questionnaire (FFQ)

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Perez Ruiz, MD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Escuela de Doctorado e Investigacion, Universidad Europea, Villaviciosa de Odón, Spain